CLINICAL TRIAL: NCT07390006
Title: Enabling Patient-Reported Outcomes Through Innovative Care Approach in Thai Older Adults Post-Acute Coronary Syndrome: A Mixed Methods Experimental Design
Brief Title: Enabling Patient-Reported Outcomes Through Innovative Care - ACS (EPIC-ACS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MURA2026/42; COA. No. MURA2026/42 (Other: Ramathibodi IRB, Mahidol University)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Coronary Syndrome/ Myocardial Infarction; Coronary Artery Disease
Keywords: Acute Coronary Syndrome; Mobile Health; Nurse-led Counseling; Patient Reported Outcome; Older Adult
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group, superiority randomized controlled trial model with two arms. Eligible participants are randomly assigned in a 1:1 ratio to either an intervention group receiving an innovative nurse-led care approach or a control group receiving usual post-acute coronary syndrome (ACS) care. Randomization occurs at the individual participant level after completion of baseline assessment. Outcomes are measured repeatedly over time to compare changes between groups during a 12-week follow-up period. The quantitative trial is complemented by a post-intervention qualitative component conducted among a subset of participants in the intervention group to further explore participant experiences.
Who Masked: Outcomes Assessor
Masking Description: This study will be a single-blind randomized controlled trial. The independent statistician, who will generate the randomization sequence, and outcome assessors will be blinded to group allocation to minimize assessment bias when collecting and analyzing patient-reported outcomes and hospital visit data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention Group - Innovative Care Approach (Experimental): Participants randomized to the intervention group will receive an innovative care approach in addition to usual post-acute coronary syndrome (ACS) care. The intervention includes a structured face-to-face education and skill-building session, provision of the Healthy Heart Booklet and motivational posters, and individualized motivational counseling focused on promoting healthy behaviors. Participants will also receive ongoing mobile health (mHealth) support delivered via the LINE application, including educational messages and motivational content to reinforce self-management behaviors. The intervention is delivered over a 12-week period to support recovery after hospital discharge and promote sustained healthy behaviors.
  Interventions: Behavioral: Innovative Care Approach
- Arm 2: Control Group - Usual Care (Active Comparator): Participants randomized to the control group will receive usual post-acute coronary syndrome (ACS) care. Usual care includes regularly scheduled follow-up visits with cardiologists at approximately 12-week intervals, medication review and adjustment as clinically indicated, and standard brief verbal education on secondary prevention behaviors, including heart-healthy diet, safe physical activity, and adherence to prescribed medication regimens provided by cardiologists and nursing staff. Participants in this group will also receive printed educational materials provided by the researcher. No additional mobile health support or structured motivational intervention will be provided.
  Interventions: Other: Usual Post-Acute Coronary Syndrome Care

INTERVENTIONS:
Behavioral: Innovative Care Approach — A nurse-led behavioral intervention including structured education, motivational counseling, and mobile health (mHealth) support delivered via the LINE application over 12 weeks.
  Arms: Arm 1: Intervention Group - Innovative Care Approach
Other: Usual Post-Acute Coronary Syndrome Care — Standard post-acute coronary syndrome care provided according to routine clinical practice.
  Arms: Arm 2: Control Group - Usual Care

SUMMARY:
This study evaluates the effectiveness of an innovative care approach that integrates face-to-face education, motivational counseling, and mobile health (mHealth) support delivered via the LINE application among Thai older adults following acute coronary syndrome (ACS) treated with percutaneous coronary intervention (PCI). The intervention aims to support post-discharge recovery by promoting healthy behaviors, improving health status, and enhancing patient satisfaction with care.

The primary objective is to assess the effect of the intervention on patient-reported outcomes, including healthy behaviors, health status, and patient satisfaction. Secondary objectives include evaluating unplanned hospital visits during a 12-week follow-up period and exploring participants' experiences, motivation, and engagement with the innovative care approach.

DETAILED DESCRIPTION:
This is a single-site, mixed-methods experimental study designed to evaluate the effectiveness of an innovative care approach among older adults following acute coronary syndrome (ACS) treated with percutaneous coronary intervention (PCI). The intervention integrates structured face-to-face education and skill-building sessions, individualized motivational counseling, and mobile health (mHealth) support delivered via the LINE application.

The quantitative component is a parallel-group, superiority randomized controlled trial with repeated measures. Eighty participants will be enrolled and randomly assigned in a 1:1 ratio to either the intervention group (innovative nurse-led care approach) or the control group (usual post-ACS care). Randomization will occur after baseline assessment using a computer-generated sequence with allocation concealment, and analyses will follow the intention-to-treat principle.

The intervention will be delivered over a 12-week period. Quantitative assessments of patient-reported outcomes will be conducted at baseline, week 8, and week 12. The qualitative component will use a post-intervention descriptive design, with in-depth interviews conducted between weeks 13 and 16 among a subset of intervention participants to explore experiences, perceived benefits, motivation, and engagement. A sequential explanatory mixed-methods approach will be used to contextualize quantitative findings with qualitative insights.

Quantitative data will be analyzed using descriptive statistics and generalized estimating equations to assess longitudinal changes over time and between groups. Unplanned hospital visits during the follow-up period will be analyzed using appropriate regression models for count data. Qualitative data will be analyzed using thematic analysis, and integration of findings will occur during interpretation.

The study has received institutional ethics approval. Written informed consent will be obtained from all participants, and confidentiality and data security will be maintained throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the quantitative phase:

1. Aged ≥ 60 years old.
2. Diagnosed with ACS and received PCI within 3-12 months.
3. Being familiar with using a smartphone or tablet with the LINE application, either personally or through a caregiver or family member.
4. No cognitive impairment assessed by the 6-Item Cognitive Function Test-Thai Version (6CIT), score less than 8.
5. Able to communicate in the Thai language by speaking, listening, reading, and writing in Thai sufficiently.
6. Voluntarily agreed to participate and has signed the informed consent form.

Inclusion Criteria for the qualitative phase:

1. Participate in the experimental group and complete the program.
2. Extreme case sampling involves selecting the top 6 highest and top 6 lowest scores for healthy behavior.
3. Willing to participate in a one-on-one in-depth interview.

Exclusion Criteria:

Exclusion Criteria for the quantitative phase:

1. Have clinical contraindications to physical exercise (i.e. unstable angina, uncontrolled arrhythmias, systolic >180 mmHg or diastolic >110 mmHg, an LVEF of less than 40%, recent major surgery within 12 weeks such as CABG, valve replacement, or orthopedic surgery), or any serious medical condition that the cardiologist considers unsafe to perform physical activity.
2. Visual or hearing impairments that cannot be adequately managed with medical devices (e.g., eyeglasses or hearing aids) and that interfere with the ability to participate in study activities or communicate effectively.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-10 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Healthy behaviors | Baseline, 8 weeks, and 12 weeks
  Healthy behaviors refer to adhering to recommended healthy lifestyle changes, mainly in diet, physical activity, medication adherence, and other relevant self-care behaviors, including avoiding smoking or second-hand smoke, air pollution, managing stress, and avoiding getting sick, especially flu infections. The Thai version of the Self-Care of Coronary Heart Disease Inventory Version 3 (SC-CHDI-V3) will be applied to measure healthy behaviors. The standardized score ranges from 0 to 100; the cut-off point scores lower than 70 indicate inadequate self-care maintenance behaviors (poor healthy behaviors); in contrast, a score of 70 or higher indicates good self-care maintenance behaviors (good healthy behaviors).
Health status | Baseline, 8 weeks, and 12 weeks
  Health status refers to treatment outcomes perceived by older participants, including symptom burden, functional status, and quality of life. Symptom burden refers to the frequency, severity, and impact of symptoms related to ACS, such as chest pain, chest tightness, or angina, while functional status is the patient's ability to perform daily activities and maintain independence, such as walking, housekeeping, and other activities. It reflects how well the patient is able to perform day-to-day activities. Quality of life indicates the overall perception of satisfaction in their life. The health status will be measured using the Seattle Angina Questionnaire (SAQ-7). The SAQ-7 score ranges from 0 - 100, with higher scores indicating less angina, fewer functional limitations, and better quality of life.
Patient satisfaction | Baseline, 12 weeks (Intervention group only)
  Patient satisfaction is the patients' level of satisfaction with the care they received, including their experiences with the innovative care approach and mHealth technology, as well as their interactions with healthcare providers. It will be measured by the Patient Satisfaction with Nurse Care Questionnaire (PSNCQ). The PSNCQ score ranges from 15 to 75; a low score indicates a lower level of satisfaction, while a higher score indicates greater satisfaction.

SECONDARY OUTCOMES:
Unplanned hospital visit | Cumulative count up to week 12
  Unplanned hospital visit refers to a situation in which an older person post-ACS needs medical care at a hospital without a prior appointment or scheduled visit, including urgent care at the emergency departments or hospital admissions. The number of unplanned emergency department visits or unplanned hospital admissions within the 12-week study period will be recorded. Data will be collected from the electronic hospital records (EHR).

OTHER OUTCOMES:
Participant Experiences With the Innovative Care Approach | Weeks 13-16
  Participant experiences regarding perceived benefits, motivation, and engagement in adhering to the innovative care approach will be explored through semi-structured in-depth interviews. Qualitative data will be analyzed using thematic analysis to provide contextual understanding of the quantitative findings.

CONTACTS AND LOCATIONS:
Overall Officials: Jamchan Prateepmanowong, PhD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Study findings will be reported in aggregate form only, in accordance with institutional review board approval and participant consent.

REFERENCES:
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Moons P, Norekval TM, Arbelo E, Borregaard B, Casadei B, Cosyns B, Cowie MR, Fitzsimons D, Fraser AG, Jaarsma T, Kirchhof P, Mauri J, Mindham R, Sanders J, Schiele F, Torbica A, Zwisler AD. Placing patient-reported outcomes at the centre of cardiovascular clinical practice: implications for quality of care and management. Eur Heart J. 2023 Sep 21;44(36):3405-3422. doi: 10.1093/eurheartj/ehad514. PMID 37606064
- [Background] Cruz-Cobo C, Bernal-Jimenez MA, Vazquez-Garcia R, Santi-Cano MJ. Effectiveness of mHealth Interventions in the Control of Lifestyle and Cardiovascular Risk Factors in Patients After a Coronary Event: Systematic Review and Meta-analysis. JMIR Mhealth Uhealth. 2022 Dec 2;10(12):e39593. doi: 10.2196/39593. PMID 36459396
- [Background] Zhu Y, Zhao Y, Wu Y. Effectiveness of mobile health applications on clinical outcomes and health behaviors in patients with coronary heart disease: A systematic review and meta-analysis. Int J Nurs Sci. 2024 Mar 10;11(2):258-275. doi: 10.1016/j.ijnss.2024.03.012. eCollection 2024 Apr. PMID 38707688
- [Background] Damluji AA, Forman DE, Wang TY, Chikwe J, Kunadian V, Rich MW, Young BA, Page RL 2nd, DeVon HA, Alexander KP; American Heart Association Cardiovascular Disease in Older Populations Committee of the Council on Clinical Cardiology and Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Radiology and Intervention; and Council on Lifestyle and Cardiometabolic Health. Management of Acute Coronary Syndrome in the Older Adult Population: A Scientific Statement From the American Heart Association. Circulation. 2023 Jan 17;147(3):e32-e62. doi: 10.1161/CIR.0000000000001112. Epub 2022 Dec 12. PMID 36503287
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654